CLINICAL TRIAL: NCT04291573
Title: Recovering Arm Function in Chronic Post-stroke Patients Using Combined HD-tDCS and Virtual Reality Therapy
Acronym: ReArm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Université Montpellier (Other); Groupement Interrégional de Recherche Clinique et d'Innovation (Other); IMT Mines Alès (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: RECHMPL19_0080; 2019-A00506-51 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2020-01-03; First posted 2020-03-02 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-04

CONDITIONS: Chronic Post Stroke Individuals
Keywords: Stroke; HD-tDCS; Virtual Reality Therapy; Physical therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HD-tDCS and Virtual Reality Therapy (Active Comparator): Patients will receive their usual rehabilitation program each day, which includes a conventional session (30min) and virtual reality therapy session (Armeo Spring) combined with real stimulation (30min) over 13 consecutive training days (3 weeks)
  Interventions: Device: HD-tDCS
- Sham stimulation and Virtual Reality Therapy (Sham Comparator): Patients will receive their usual rehabilitation program each day, which includes a conventional session (30min) and virtual reality therapy session (Armeo Spring) combined with Sham stimulation (30min) over 13 consecutive training days (3 weeks)
  Interventions: Device: Sham HD-tDCS

INTERVENTIONS:
Device: HD-tDCS — Real stimulation (2mA, 20min) with anode on C3/C4 of the lesioned hemisphere and 4 return electrodes ~4cm away
  Other Names: Starstim8 (Neuroelectrics, Spain)
  Arms: HD-tDCS and Virtual Reality Therapy
Device: Sham HD-tDCS — Sham stimulation (2mA, ramp up and down phases of 30s) with anode on C3/C4 of the lesioned hemisphere and 4 return electrodes ~4cm away
  Other Names: Starstim8 (Neuroelectrics, Spain)
  Arms: Sham stimulation and Virtual Reality Therapy

SUMMARY:
The study aims to determine the added value of combining high-definition transcranial direct current stimulation (HD-tDCS) in a rehabilitation program based on virtual reality therapy (VRT) to potentiate the effects on neuroplasticity and further improve functional recovery of the arm in chronic stroke patients.

DETAILED DESCRIPTION:
Stroke remains the leading cause of acquired disability in France. Moreover, even after the first 3 months of intense arm rehabilitation, 80% of chronic stroke patients don't use their paretic arm in activities of daily living.

To this day, despite notable developments, techniques of rehabilitation of the arm for chronic stroke patients are still insufficient. In this context, two promising stroke rehabilitation techniques are to be considered:

* Virtual reality-based systems provide specific, intensive, repetitive and motivational therapy with real-time feedback of movement and performance which can promote activity-dependent brain neuroplasticity, and therefore functional arm recovery. Thus, virtual reality therapy (VRT), in addition to usual rehabilitation, would improve the function of the arm more effectively as well as daily activities.
* Non-invasive transcranial direct current stimulation (tDCS) uses constant low intensity (2 mA) continuous electrical currents to modulate the excitability of cortical neurons. Because of its greater focality of neuromodulatory effect that promotes brain neuroplasticity, anodal HD-tDCS to the lesioned hemisphere can improve functional arm recovery after a stroke. In addition, the combined use of the HD-tDCS with a rehabilitation modality, such as constraint induced movement therapy, would potentiate the combined effects of both techniques.

Therefore, the investigators hypothesize that the combination of HD-tDCS in a rehabilitation program based on VRT would potentiate the effects on neuroplasticity and would further improve functional recovery of the paretic arm in chronic stroke patients

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 to 90
* Patient with more than 3 months of a first cerebrovascular accident whatever the aetiology
* Patient with paresis of the upper extremity (FM-UE ≥ 15)

Exclusion Criteria:

* Failure to collect written informed consent after a period of reflection
* Not be affiliated with a French social security scheme or beneficiary of such a scheme
* Major deficit of the upper extremity (FM-UE <15)
* History of epilepsy
* Presence of a pacemaker or a metallic object implanted in the head
* Pregnant or lactating
* Severe neglect or attention deficit disorder (omission of more than 15 bells in the Bell's test)
* Severe cognitive impairment (Mini Mental Score <24)
* Aphasia with impairment of understanding (Boston Aphasia Quotient <4/5)
* Under guardianship or curatorship
* Protected by law

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Change in Functional Motor capacity of the upper extremity | Change from Baseline at Day 21(after intervention) and 3 months after day 21
  Arm functional capacity assessed by the Wolf Motor Function Test (WMFT) (0-75, where higher scores mean better arm functional capacity)
Change in Functional Motor capacity of the upper extremity | Change from Day 21 at 3 months (retention)
  Arm functional capacity assessed by the Wolf Motor Function Test (WMFT) (0-75, where higher scores mean better arm functional capacity)
Change in Motor deficit of the upper extremity | Change from Baseline at Day 21 (after intervention) and 3 months after day 21
  Measured by the Fugl-Meyer Upper Extremity (FMUE) score (0-66, where higher scores mean a better recovery)
Change in Motor deficit of the upper extremity | Change from Day 21 at 3 months (retention)
  Measured by the Fugl-Meyer Upper Extremity (FMUE) score (0-66, where higher scores mean a better recovery)
Change in Hand dexterity | Change in Baseline at Day 21 (after intervention) and 3 months after day 21
  Measured by the Box and Block Test (BBT) score (greater number of blocks moved in 1minute means better hand dexterity)
Change in Hand dexterity | Change in Day21 at 3 months (retention)
  Measured by the Box and Block Test (BBT) score (greater number of blocks moved in 1minute means better hand dexterity)

SECONDARY OUTCOMES:
Change in Non-use of the paretic upper extremity | Change from Baseline at Day 21 (after intervention) and 3 months after day 21
  Measured by the Proximal Arm Non-Use (PANU) score during an arm reaching task (0-100 where higher scores mean a worse outcome)
Change in Non-use of the paretic upper extremity | Change from Day 21 at 3 months (retention)
  Measured by the Proximal Arm Non-Use (PANU) score during an arm reaching task (0-100 where higher scores mean a worse outcome)
Change in Activities of daily living | Change from Baseline at Day 21 (after intervention) and 3 months after day 21
  Measured by the Barthel Index (0-100 where higher scores mean a better outcome)
Change in Activities of daily living | Change from Day 21 at 3 months (retention)
  Measured by the Barthel Index (0-100 where higher scores mean a better outcome)
The use of the paretic upper extremity in activities of daily living | Change from Baseline at Post (10 days after the intervention), and Post 3 months (10 days at 3 months post intervention)
  Measured by the magnitude and ratio of arm movements over a 10-day period from wrist worn accelerometers on each arm
The use of each upper extremity in activities of daily living | Change from Post at Post 3 months (retention)
  Measured by the magnitude and ratio of arm movements over a 10-day period from wrist worn accelerometers on each arm

OTHER OUTCOMES:
Change in Interhemispheric Sensorimotor cortex haemodynamics (functional near-infrared spectroscopy-fNIRS) | Change from Baseline at Day 21 (after intervention)
  Measured by the magnitude and ratio of the concentration of oxygenated haemoglobin in the ipsilesional and contralesional sensorimotor cortex at rest and during arm movements
Change in Interhemispheric Sensorimotor cortex haemodynamics (functional near-infrared spectroscopy-fNIRS) | Change from Day 21 at 3 months (retention)
  Measured by the magnitude and ratio of the concentration of oxygenated haemoglobin in the ipsilesional and contralesional sensorimotor cortex at rest and during arm movements
Change in Interhemispheric Sensorimotor cortex neural oscillations (Electroencephalography- EEG) | Change from Baseline at Day 21 (after intervention)
  Measured by the magnitude and ratio of alpha/beta frequency power in the ipsilesional and contralesional sensorimotor cortex at rest and during arm movements
Change in Interhemispheric Sensorimotor cortex neural oscillations (Electroencephalography- EEG) | Change from Day 21 at 3 months (retention)
  Measured by the magnitude and ratio of alpha/beta frequency power in the ipsilesional and contralesional sensorimotor cortex at rest and during arm movements

CONTACTS AND LOCATIONS:
Overall Officials: Karima KA Bakhti, PhD, Principal Investigator — Montpellier hospital Lapeyronie
Locations (1):
- Montpellier hospital Lapeyronie, Montpellier, France

IPD SHARING:
Plan to Share IPD: Yes
Data available upon request through a data access

REFERENCES:
- [Background] Levin MF, Weiss PL, Keshner EA. Emergence of virtual reality as a tool for upper limb rehabilitation: incorporation of motor control and motor learning principles. Phys Ther. 2015 Mar;95(3):415-25. doi: 10.2522/ptj.20130579. Epub 2014 Sep 11. PMID 25212522
- [Background] Laffont I, Bakhti K, Coroian F, van Dokkum L, Mottet D, Schweighofer N, Froger J. Innovative technologies applied to sensorimotor rehabilitation after stroke. Ann Phys Rehabil Med. 2014 Nov;57(8):543-551. doi: 10.1016/j.rehab.2014.08.007. Epub 2014 Aug 26. PMID 25261273
- [Background] Laver KE, Lange B, George S, Deutsch JE, Saposnik G, Crotty M. Virtual reality for stroke rehabilitation. Cochrane Database Syst Rev. 2017 Nov 20;11(11):CD008349. doi: 10.1002/14651858.CD008349.pub4. PMID 29156493
- [Background] Polania R, Nitsche MA, Ruff CC. Studying and modifying brain function with non-invasive brain stimulation. Nat Neurosci. 2018 Feb;21(2):174-187. doi: 10.1038/s41593-017-0054-4. Epub 2018 Jan 8. PMID 29311747
- [Background] Bikson M, Grossman P, Thomas C, Zannou AL, Jiang J, Adnan T, Mourdoukoutas AP, Kronberg G, Truong D, Boggio P, Brunoni AR, Charvet L, Fregni F, Fritsch B, Gillick B, Hamilton RH, Hampstead BM, Jankord R, Kirton A, Knotkova H, Liebetanz D, Liu A, Loo C, Nitsche MA, Reis J, Richardson JD, Rotenberg A, Turkeltaub PE, Woods AJ. Safety of Transcranial Direct Current Stimulation: Evidence Based Update 2016. Brain Stimul. 2016 Sep-Oct;9(5):641-661. doi: 10.1016/j.brs.2016.06.004. Epub 2016 Jun 15. PMID 27372845
- [Background] Chhatbar PY, Chen R, Deardorff R, Dellenbach B, Kautz SA, George MS, Feng W. Safety and tolerability of transcranial direct current stimulation to stroke patients - A phase I current escalation study. Brain Stimul. 2017 May-Jun;10(3):553-559. doi: 10.1016/j.brs.2017.02.007. Epub 2017 Feb 27. PMID 28279641
- [Background] Floel A. tDCS-enhanced motor and cognitive function in neurological diseases. Neuroimage. 2014 Jan 15;85 Pt 3:934-47. doi: 10.1016/j.neuroimage.2013.05.098. Epub 2013 May 30. PMID 23727025
- [Background] Teo WP, Muthalib M, Yamin S, Hendy AM, Bramstedt K, Kotsopoulos E, Perrey S, Ayaz H. Does a Combination of Virtual Reality, Neuromodulation and Neuroimaging Provide a Comprehensive Platform for Neurorehabilitation? - A Narrative Review of the Literature. Front Hum Neurosci. 2016 Jun 24;10:284. doi: 10.3389/fnhum.2016.00284. eCollection 2016. PMID 27445739
- [Background] Allman C, Amadi U, Winkler AM, Wilkins L, Filippini N, Kischka U, Stagg CJ, Johansen-Berg H. Ipsilesional anodal tDCS enhances the functional benefits of rehabilitation in patients after stroke. Sci Transl Med. 2016 Mar 16;8(330):330re1. doi: 10.1126/scitranslmed.aad5651. Epub 2016 Mar 16. PMID 27089207
- [Background] Bakhti KKA, Laffont I, Muthalib M, Froger J, Mottet D. Kinect-based assessment of proximal arm non-use after a stroke. J Neuroeng Rehabil. 2018 Nov 14;15(1):104. doi: 10.1186/s12984-018-0451-2. PMID 30428896
- [Background] Chhatbar PY, Ramakrishnan V, Kautz S, George MS, Adams RJ, Feng W. Transcranial Direct Current Stimulation Post-Stroke Upper Extremity Motor Recovery Studies Exhibit a Dose-Response Relationship. Brain Stimul. 2016 Jan-Feb;9(1):16-26. doi: 10.1016/j.brs.2015.09.002. Epub 2015 Sep 7. PMID 26433609
- [Background] Figlewski K, Blicher JU, Mortensen J, Severinsen KE, Nielsen JF, Andersen H. Transcranial Direct Current Stimulation Potentiates Improvements in Functional Ability in Patients With Chronic Stroke Receiving Constraint-Induced Movement Therapy. Stroke. 2017 Jan;48(1):229-232. doi: 10.1161/STROKEAHA.116.014988. Epub 2016 Nov 29. PMID 27899754
- [Derived] Dusfour G, Mottet D, Muthalib M, Laffont I, Bakhti K. Comparison of wrist actimetry variables of paretic upper limb use in post stroke patients for ecological monitoring. J Neuroeng Rehabil. 2023 Apr 27;20(1):52. doi: 10.1186/s12984-023-01167-y. PMID 37106460
- [Derived] Muller CO, Muthalib M, Mottet D, Perrey S, Dray G, Delorme M, Duflos C, Froger J, Xu B, Faity G, Pla S, Jean P, Laffont I, Bakhti KKA. Recovering arm function in chronic stroke patients using combined anodal HD-tDCS and virtual reality therapy (ReArm): a study protocol for a randomized controlled trial. Trials. 2021 Oct 26;22(1):747. doi: 10.1186/s13063-021-05689-5. PMID 34702317